CLINICAL TRIAL: NCT04727463
Title: Obstetric Fecal Incontinence Treatment Registry
Status: Completed | Type: Observational
Sponsor: Hospital San Carlos, Madrid (Other)
Responsible Party: Principal Investigator, Carlos Cerdán Santacruz, Principal Investigator, Hospital San Carlos, Madrid
Other Study IDs: 17/100-E
Record Dates: First submitted 2020-12-16; First posted 2021-01-27 (Actual); Last update posted 2021-01-27 (Actual); Status verified 2021-01

CONDITIONS: Fecal Incontinence
MeSH Terms: conditions — Fecal Incontinence | interventions — Sphincterotomy, Transduodenal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Sphincteroplasty — Overlapping sphincteroplasty

SUMMARY:
INTRODUCTION Anal Incontinence (AI) is a loose of voluntary control for bowel movements, with recurrent leaking of flatus, liquid or solid stools.

AI is a frecuent pathology. Prevalence is similar among men and women. AI´s ethiology is quite variable. Nevertheless, the most frecuent one is sphinteric injuries, obstetric, traumatic or secondary to anal surgery.

Conservative measures have to be iniciated and they are essential for every patient.

If a sphincteric injury exists, several choices of surgical treatment exist. The long term results obtained with sphincteroplasty, with a uniform surgical technique, follow up and complementing with other therapeutic options, has been considered interesting to analyze.

HYPOTHESIS Sphincteroplasty with the adoption of the appropriate complementary treatments, provides satisfactory results in the very long term, and should be considered as the procedure of choice in patients with Anal Incontinence.

OBJECTIVES

* Analyze the very long term results obtained with Sphincteroplasty as surgical technique for treatment of severe anal incontinence.
* Evaluate the results of the different types of surgical repair performed, according to the CCIS Score (Wexner Score).
* Evaluate the importance of patient follow-up and incorporation of complementary treatments.
* Establish patient´s satisfaction with the procedure after a long term follow up period after the intervention.

DETAILED DESCRIPTION:
MATERIAL AND METHODS

PATIENTS AND METHOD A retrospective Cohort study was designed, based on a prospectively maintained database, including every consecutive patient operated on severe AI secondary to sphincteric injury with sphincterolplasty, between January 1985 and December 2013.

Every operations were performed by the same surgeon in two centers, Hospital Clinico San Carlos and Santa Elena Clinic, both in Madrid.

INCLUSION CRITERIA Every patients, without limitation of gender or age, with any kind of sphincteric lesion susceptible of surgical repair, presenting with AI and severe impairment in quality of life, after following a conservative treatment and unsatisfactory results.

EXCLUSION CRITERIA There are not exclusion criteria except non-fitting inclusion criteria.

INDEPENDENT VARIABLES EVALUATED The independent variables considered for the analysis are age, gender, etiologic factors, impact on daily life measured with the Wexner et al Score (CCIS), diagnostic tests used, type of surgical intervention performed, obtained results and long term satisfaction reached with the procedure.

A.- PREOPERATIVE EVALUATION

1. - Exhaustive anamnesis to determine the severity of AI using the Wexner Score (CCIS).
2. - Anal and perineal exploration to determine the extension of sphincteric lesion and exclude other possible pathologies.
3. - Complementary tests, mainly ano-rectal Manometry and Endo-Anal Ultrasound. Other tests chosen selectively in certain cases.

B.- OPERATIVE DETAILS All patients underwent antegrade mechanic colon cleansing and antibiotic and thromboembolic prophylaxis. Under general or spinal anesthesia the patient is fixed in lithotomy position, the rectum is irrigated and a meticulous cleansing of the vagina is done.

Skin incision of a sufficient size is done to facilitate the appropriate dissection and freedom of the sphincter endings.

If it was a "clear" lesion of the external Sphincter, a tensión-free overlapping with absorbable 2/0 material is performed. If accompanying internal anal sphincter lesion was found, a suturing or plication of the anterior rectal wall, including internal anal sphincter fibres was done. Finally, when a levatorplasty is also going to be associated, the whole procedure includes the plication of the internal anal sphincter, levatorplasty by the midline plication of the pubo-rectalis muscle with two or three stitches and, at the end, the external anal sphincter overlapping sphincteroplasty.

When any other ano-rectal disorder was also identified it was simultaneously repaired.

C.- POSTOPERATIVE FOLLOW-UP All the patients are exhaustively followed in the clinic for postoperative sphincteric function assesing and individualized counseling depending on their progress, varying from dietetic and farmacological advice, biofeedback prescription, or even the indication of further surgical treatments when necessary.

It was stablished a follow-up visit every six months during the first three postopeative years, and then anual visits until the fifth postoperative year. From this point every year a in-person or telephone control was kept, selected by each patient based on personal preferences.

If an improvable sphincter anal function is detected during follow up, although no heavily impacting on quality of life, prescription of biofeedback therapy was done. If a more significative impact was determined, biofeedback during the first years and posterior tibial nerve stimulation (PTNS) or SNS the last years.

Criteria for the different options prescription was based on an individualized evaluation of quality of life, advantages, disadvantages and always centered in benefiting the patient.

D.- PERSONAL INTERVIEW / DEFINITE EVALUATION: LAST FOLLOW-UP For the completion of this study, it was decided to carry out simple assessments based on easy to answer questions that reflected as accurately as possible the situation of each patient, discarding for this reason the use of any of the quality of life scales.

Similar parameters to those used in other studies have been used, both through direct or telephone interview conducted from September through November 2015. A total of 105 patients who had undergone surgery in the past were interviewed and this was considered as "the last control".

Throughout this interview the following infomation was recruited:

1. - CCIS.
2. - Questions focusing in determine level of satisfaction:

   1. - Browning-Parks´ Scale
   2. - Clinic Score.
   3. - Visual Analogic Scale (VAS).
   4. - Subjective Situation after Surgery.
   5. - Would you take the operation again?
   6. - Would you recomend the operation to any friendo r relative?

STATISTICAL METHOD Statistical Analysis Qualitative variables are presented by their frecuency distribution. Quantitative variables are summarized in their mean and standard deviation (SD) or median and interquartile range (IQR) in cases of asymmetry.

Variation of quantitative variables was studied with the T of Student test for paired data and analysis of variance for repeated measures (ANOVA), correcting significance level with Bonferroni´s test. Mean absolute effects and their 95% confidence intervals (95% CI) were estimated. We adjusted covariance models to evaluate the variables related to the final Wexner score adjusted for the initial values.

In all cases, the distribution of the variable was checked against the theoretical models and the variance homogeneity hypothesis was contrasted.

In every hypothesis contrasts, the null hypothesis was rejected with a type I error or an α error less than 0.05.

The statistical package used for the analysis was SPSS for Windows version 20.0.

ETHICAL ASPECTS AND CONFIDENTIALITY Ethical and legal aspects This work respects ethical and legal rules applicable to this type of studies and follows the rules of good clinical practice in its realization, according to the Law 14/2007 of the 4th of July of Biomedical Research.

Approval was requested from the Clinical Research Ethics Committee of the Hospital Clínico San Carlos to carry out the study. This Committee granted the authorization as well as, where appropriate, the publication of the results.

Confidentiality All the findings obtained in this investigation will be kept confidential, guaranteeing compliance with the principles established in the Organic Law of Protection of Personal Data 15/1999 of December 13 and facilitating the exercise of rights of access, rectification, cancellation and opposition.

In case of publication of the results of the study, the identity of the patients will not be revealed.

Conflict of interests Neither the PhD student, nor the Directors, nor any of the surgeons who have participated in the care of patients, present any conflict of interest.

ELIGIBILITY:
Inclusion Criteria:

* Any person with kind of sphincteric lesion susceptible of surgical repair.
* Presenting with Anal Incontinence and severe impairment in quality of life.
* Unsatisfactory results after following a conservative treatment.

Exclusion Criteria:

* Not exclusion criteria except non-fitting inclusion criteria.

Ages: 16 Years to 84 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: 113 women (94.2%) and 7 men (5.8%), aged between 16 and 84 years old.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2020-12-16 (Actual); Primary Completion 2020-12-16 (Actual); Study Completion 2020-12-16 (Actual)

PRIMARY OUTCOMES:
Cleveland Clinic Incontinence Score | Up to 5 years
  Retrospective cohort Study

CONTACTS AND LOCATIONS:
Locations (1):
- Carlos Cerdán, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No